CLINICAL TRIAL: NCT01265030
Title: A Pilot Study Evaluating the Use of mTor Inhibitor Sirolimus in Children and Young Adults With Desmoid-Type Fibromatosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MaineHealth (Other)
Collaborators: Desmoid Tumor Research Foundation (Other); Pfizer (Industry)
Responsible Party: Principal Investigator, Aaron Weiss, Principal Investigator, MaineHealth
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-491-B; 44574 (Other Grant/Funding Number: Desmoid Tumor Research Foundation)
Record Dates: First submitted 2010-12-06; First posted 2010-12-22 (Estimated); Results first posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Desmoid Tumor
Keywords: Desmoid Tumor; Sirolimus; Surgically-Resectable Desmoid Tumor
MeSH Terms: conditions — Desmoid Tumors | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | US Export: Yes

ARMS (1):
- Sirolimus (Experimental): Preoperative sirolimus:
  * loading dose of 12 milligrams/meter2; Per Os (PO), by mouth day 1 (Max dose 12 milligram)
  * starting 24 hours after the initial loading dose, subjects will receive a dose of 4 milligram/meters2 daily; Per Os (PO), by mouth days 2 through 28
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — * Loading dose of 12 milligrams/meter2; Per Os (PO), by mouth day 1 (Max dose 12 milligrams)
  * Starting 24 hours after the initial loading dose, patients will receive a dose of 4 milligrams/meter2 daily; Per Os (PO), by mouth days 2 through 28 (Max dose 4 milligram/day)
  Other Names: Rapamune®; Rapamycin

SUMMARY:
Desmoid-type fibromatosis (or desmoid tumor) represents an intermediate grade neoplasm with a striking predilection for locally invasive growth and recurrence following resection. It occurs in children as well as young adults. As a typically localized disease, the historical standard of care for treatment has been surgical resection, with or without ionizing radiation. In some cases where surgical resection or radiation is not feasible, chemotherapy has been used. Two clinical trials conducted in the Pediatric Oncology Group (POG) and the Children's Oncology Group (COG) evaluated the role for either low intensity or non-cytotoxic chemotherapy for children with desmoid tumor that is not amenable to standard therapy. These were largely empirical treatment strategies or based on somewhat anecdotal observations. By better understanding desmoid tumor biology, even more effective therapy targeting a particular protein that is central to the disease can be developed.

Desmoid tumor is well-known to be associated with deregulation of the Adenomatous Polyposis Cell/beta-catenin (APC/β-catenin pathway). This is true of familial cases associated with Gardner's Syndrome and also in sporadic desmoid tumor, nearly all of which display histological or molecular evidence of Adenomatous Polyposis Cell/beta-catenin (APC β-catenin) pathway activation (Alman et al., 1997; Lips et al., 2009). Several new pieces of evidence support the concept that deregulation of the mammalian target of rapamycin (mTOR) cell proliferation/survival pathway may play an important role in tumor biology when the APC/β-catenin pathway is disrupted. Sirolimus, a drug that inhibits mammalian target of rapamycin (mTOR), is currently being evaluated as an anti-cancer agent in a variety of tumor types, but it has not been previously studied in desmoid tumor.

The investigators are conducting this pilot study to begin to explore whether mTOR inhibition may be beneficial for children and young adults with desmoid tumor.

DETAILED DESCRIPTION:
We propose a translational research project that will directly test the hypothesis that mTOR is active in desmoid tumor in children and young adults. Activity will be assessed by clinical and histological studies following a course of pre-operative chemotherapy using sirolimus. Clinical response will be measured using validated pain assessment scales because desmoid tumor size is unlikely to change during the course of pre-operative chemotherapy in this study. Histological response will be based on quantifying the phosphorylation of following mTOR targets: thr389p-p70S6K, p-4E-BP1, and ser473p-AKT.

ELIGIBILITY:
Inclusion Criteria:

* Must be less than 30 years of age at time of original diagnosis
* Must have biopsy-proven desmoid tumor (or aggressive fibromatosis). For patients with recurrent disease, a biopsy is not required at the time of recurrence
* Patients known to have germ-line adenomatous polyposis coli (APC) mutations or clinical manifestations of Familial Adenomatous Polyposis(FAP)/Gardner's syndrome can be included
* Patients must have surgery planned to remove the desmoid tumor and either:

  * the desmoid tumor has already recurred after a prior surgery or
  * the newly diagnosed and/or previously unresected disease is judged to be at high risk for recurrence due to its size (>5 centimeters) or location at an anatomic site making it unlikely to be resected with negative margins (eg. adjacent to neurovascular structures)
* There must be a commitment by the surgical team to resect the primary tumor within 3 days following the 4 weeks of sirolimus unless the clinical situation at the time of resection suggests that these interventions are not in the patient's best interest
* Concomitant medication restrictions:

  * Patients may have received prior chemotherapy (excluding prior mTOR inhibitors)
  * Use of steroids for non-tumor indications (for example: asthma or severe allergic reaction) is permitted
* Patients must have a Karnofsky performance status of greater than or equal to 50 for patients older than 16 years of age or Lansky performance status of greater than or equal to 50 for patients less than or equal to 16 years of age.
* Patients must have a life expectancy of greater than or equal to 8 weeks.
* Patients must have recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study

  * Myelosuppressive chemotherapy: Must not have received within 2 weeks of entry onto this study (4 weeks if prior nitrosourea)
  * Biologic (anti-neoplastic agent): at least 7 days since the completion of therapy with a biological agent
  * Stem Cell Transplant (SCT): No evidence of active graft versus host disease. For allogeneic SCT, greater than or equal to 6 months must have elapsed.
* Patients must be able to consume oral medication in the form of tablets or solution
* Patients must have normal laboratory values as defined below:

  * Creatinine clearance or radioisotope Glomerular Filtration Rate ≥ 70millileters/minute/1.73 meters2 or a normal serum creatinine based on age/gender
* Hepatic: Adequate liver function is defined as:

  * Total bilirubin less than or equal to 1.5 x upper limit of normal (ULN)for age, and
  * Serum glutamic pyruvic transaminase (SGPT) less than or equal to 2.5 x upper limit normal (ULN) for age
* Hematologic function: Adequate bone marrow function is defined as:

  * Absolute Neutrophil Count (ANC) greater than or equal to 1 x 10 to the ninth/Liter
  * Hemoglobin greater than or equal to 10 gram/deciliter
  * Platelet count greater than or equal to 100 x 10 to the ninth/Liter
* Female patients must have a negative pregnancy test
* Female patients who are lactating must agree to stop breast-feeding
* Sexually active patients of childbearing potential must agree to use effective contraception
* Patients must be able to cooperate fully with all planned protocol therapy
* Signed informed consent MUST be obtained from patient or parent/legal guardian (if patient is less than 18 years of age). Consent must be signed prior to any study procedures and study entry

Exclusion Criteria:

* Patients with other fibroblastic lesions or other fibromatoses are NOT eligible.
* Concomitant medication restrictions

  * Patients may NOT have received prior mTor inhibitors
  * Growth factor(s): Must not have received within 1 week of entry onto this study.
* Patients must not be known to be Human Immunodeficiency Virus positive. Testing for Human Immunodeficiency Virus is not mandatory.
* Patients must not be taking medicines known to influence sirolimus metabolism

Max Age: 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2021-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron R Weiss, DO, Principal Investigator — MaineHealth
Locations (8):
- United States (8):
  - UCLA Medical Center, Los Angeles, California
  - Rady Children's Hospital, San Diego, California
  - University of Florida College of Medicine, Gainesville, Florida
  - Maine Medical Center, Portland, Maine
  - University of Minnesota, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Seattle Children's Hospital, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Sirolimus: Preoperative sirolimus:
  * loading dose of 12 milligrams/meter2; Per Os (PO), by mouth day 1 (Max dose 12 milligram)
  * starting 24 hours after the initial loading dose, subjects will receive a dose of 4 milligram/meters2 daily; Per Os (PO), by mouth days 2 through 28
  Sirolimus: -Loading dose of 12 milligrams/meter2; Per Os (PO), by mouth day 1 (Max dose 12 milligrams)
  -Starting 24 hours after the initial loading dose, patients will receive a dose of 4 milligrams/meter2 daily; Per Os (PO), by mouth days 2 through 28 (Max dose 4 milligram/day)
Period: Overall Study
Arm/Group | Sirolimus
Started (Goal enrollment of 15 subjects) | 9
Completed | 9 (9 of anticipated 15 patients accrued)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sirolimus
Number analyzed (Participants) | 9
Age, Continuous [Median (Full Range); unit: years] | 15 [5 to 28]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Immunohistochemical Immunoreactive Score Results After 4 Weeks of Sirolimus Compared to Control Specimens
Description: Changes to the mTOR pathway were determined using an immunohistochemical immunoreactive score (IRS). The components of the IRS for each phosphoprotein (p4EPB and pS706K) are as follows: the percentage of positive cells were scored as: 0 (0%); 1 (<10%); 2 (11-50%); 3 (51-80%); 4(>80%). The staining intensity were scored as: 0 (negative), 1 (weak), 2 (moderate), and 3 (strong). To derive the IRS, the percentage of positive cells and staining intensity were multiplied together, resulting in a value from 0 to 12. The score for patients after 4 weeks of sirolimus was compared to a group of control desmoid tumor samples from the UCLA tumor bank (n=68). Lower scores for patients following 4 weeks of sirolimus compared to control sample scores indicate a better outcome.
Time Frame: 4 weeks
Population: The 9 patients who were treated with sirolimus were compared to a group of control desmoid tumor samples from the UCLA tumor bank (n=68); no identifiable baseline or adverse event data were collected or available from participants who contributed control tumor samples due to anonymization.
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Immunoreactive Score Results of p4EPB After 4 Weeks of Sirolimus for the Study Patients: The mean immunohistochemical immunoreactive score (IRS) of the phosphoprotein p4EPB for the study patients following 4 weeks of sirolimus is provided.
- Immunoreactive Score Results of pS706K After 4 Weeks of Sirolimus for the Study Patients: The mean immunohistochemical immunoreactive score (IRS) of the phosphoprotein pS706K for the study patients following 4 weeks of sirolimus is presented.
- Immunoreactive Score Results of p4EPB for the Control Tumors: The mean immunohistochemical immunoreactive score (IRS) of the phosphoprotein p4EPB for the control tumor samples is presented.
- Immunoreactive Score Results of pS706K for the Control Tumors: The mean immunohistochemical immunoreactive score (IRS) of the phosphoprotein pS706K for the control tumor samples is presented.
Arm/Group | Immunoreactive Score Results of p4EPB After 4 Weeks of Sirolimus for the Study Patients | Immunoreactive Score Results of pS706K After 4 Weeks of Sirolimus for the Study Patients | Immunoreactive Score Results of p4EPB for the Control Tumors | Immunoreactive Score Results of pS706K for the Control Tumors
Number analyzed (Participants) | 9 | 9 | 68 | 68
score on a scale | 5.22 [1 to 12] | 7.44 [0 to 12] | 4.47 [0 to 12] | 9.39 [0 to 12]
Statistical Analysis 1: Comparison: Immunoreactive Score Results of p4EPB After 4 Weeks of Sirolimus for the Study Patients; Test type: Superiority; p = 0.63, t-test, 2 sided; Mean Difference (Net) = 0.75, 95% CI 2-sided [-2.54 to 4.04]
Statistical Analysis 2: Comparison: Immunoreactive Score Results of pS706K After 4 Weeks of Sirolimus for the Study Patients; Test type: Superiority; p = 0.31, t-test, 2 sided; Mean Difference (Net) = -1.95, 95% CI 2-sided [-6.08 to 2.19]

2. Secondary Outcome: Pain Levels After 4 Weeks of Sirolimus
Description: Pain assessments were performed using the validated numeric (age ≥ 10 years) and Wong-Baker FACES (≥3 and < 10 years) pain rating scales at specified study time points including baseline, at week 1 and after 4 weeks of treatment (just prior to surgery). Both pain scales range from a value of 0 to 10 with 0 being equal to no pain and 10 being equal to the worst pain. The median pain score and pain score range for study participants at Week 1 and Prior to Surgery (Week 4) timepoints are provided. Lower pain scale values (median and upper limit of the range) at the Prior to Surrgery timepoint are considered a better outcome.
Time Frame: 4 weeks
Population: Pain scores were obtained weekly throughout the 4 week study period in all participants
Measure: Median (Full Range); unit: score on a scale
Groups:
- Week 1; Prior to Surgery: Validated pain assessment measures, using the numeric (>=10 years of age) and Wong-Baker FACES (< 10 years of age) scales were collected at specific study time points. A positive response will be associated with an improvement of ≥ 50% from baseline after 4 weeks (prior to surgery). A negative response will be associated with any worsening from baseline after 4 weeks. A stable response will be any other result.
Arm/Group | Week 1 | Prior to Surgery
Number analyzed (Participants) | 9 | 9
score on a scale | 1 [0 to 3] | 0 [0 to 3]
Statistical Analysis 1: Comparison: Week 1 vs Prior to Surgery; The mean difference in pain score at week 1 and before surgery; Test type: Superiority; p = 0.68, t-test, 2 sided; Mean Difference (Net) = 0.063, 95% CI 2-sided [-.286 to 0.411]

3. Secondary Outcome: Number of Participants Without Tumor Recurrence
Description: We evaluated the number of study participants whose tumor did not recur by 3 years from the date of surgery.
Time Frame: 3 years from the end of therapy, a total duration of 3 years and 4 weeks
Population: All trial participants
Measure: Count of Participants; unit: Participants
Groups:
- Study Patients: Patients will be followed for recurrence post-surgery
Arm/Group | Study Patients
Number analyzed (Participants) | 9
Participants | 5

4. Secondary Outcome: Number of Participants With Grade 3 or Higher Toxicity Per CTCAE Definitions
Description: The safety and tolerability of patients receiving sirolimus was evaluated using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 grading criteria. All reported grades of toxicity (1-5) were collected.
Time Frame: 4 weeks
Population: All trial participants
Measure: Count of Participants; unit: Participants
Groups:
- Safety: Number of study subjects with Grade 3 or higher toxicity per CTCAE definitions
Arm/Group | Safety
Number analyzed (Participants) | 9
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of treatment (4 weeks).
Arm/Group | Sirolimus
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 7/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus (N=9)
Headache (Nervous system disorders) | 2 (2)
Fatigue (General disorders) | 2 (2)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Weight loss (Investigations) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 5 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 3 (3)
Neutrophil count decreased (Investigations) | 2 (2)
Creatinine increased (Investigations) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Hypotension (Vascular disorders) | 4 (4)
Platelet count decreased (Investigations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Sinus pain (Nervous system disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Facial pain (General disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Flu like symptoms (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-19): https://cdn.clinicaltrials.gov/large-docs/30/NCT01265030/Prot_SAP_000.pdf